CLINICAL TRIAL: NCT04156061
Title: Effect of the SCOT-HEART 2 Trial on Lifestyle and Risk Factor Modification.
Brief Title: Effect of the SCOT-HEART 2 Trial on Lifestyle.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AC19113
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Primary Prevention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASSIGN score (No Intervention): The baseline assessment will be completed on the same day as consent is gained. Every patients will complete a comprehensive assessment including questionnaires and objective assessments.
  Patients randomised to standard care with ASSIGN score alone (n=200) will be invited back approximately 6 months after baseline assessment. The detailed questionnaire, breath test, blood pressure monitoring, and 2-week activity monitor will be repeated. Bloods will be retaken to look at change in lipid levels and HbA1c where appropriate - no more than 30mls will be required.
- CTCA - visual report (Active Comparator): Those in the CTCA group will be further randomised into review with or without CT images.
  The review WITH images (VISUAL REPORT N=100) group will have results delivered by the principal investigator (a trained Cardiology Registrar) to ensure a standardised approach to relaying information. These results will be preliminary and focused only on whether the patient has evidence of coronary disease or not. A full report describing the extent of coronary disease, other cardiac problems and incidental findings will follow as per the SCOT-HEART-2 protocol. Patients will be made aware that the presented findings are a focused preliminary report and that a more detailed formal report will follow.
  Interventions: Other: Delivery of CT scan results
- CTCA - verbal report (Active Comparator): The baseline assessment will be completed on the same day as consent is gained. Every patients will complete a comprehensive assessment including questionnaires and objective assessments.
  Those in the CTCA group will be further randomised into review with or without CT images.
  The review WITHOUT images (VERBAL REPORT N=100) group will have results delivered by the principal investigator (a trained Cardiology Registrar) to ensure a standardised approach to relaying information. These results will be preliminary and focused only on whether the patient has evidence of coronary disease or not. A full report describing the extent of coronary disease, other cardiac problems and incidental findings will follow as per the SCOT-HEART-2 protocol. Patients will be made aware that the presented findings are a focused preliminary report and that a more detailed formal report will follow.
  Interventions: Other: Delivery of CT scan results

INTERVENTIONS:
Other: Delivery of CT scan results — Method of results delivery - verbal or visual.
  Arms: CTCA - verbal report; CTCA - visual report

SUMMARY:
This study will recruit 400 participants who are taking part in the Computed Tomography Coronary Angiography for the Prevention of Myocardial Infarction (SCOT-HEART 2) trial. The investigator will assess diet, activity and habits at the start of the study and 6 months later. This will help us understand the effects taking part in the study may have on lifestyle. In addition, for participants who have CT scans, the investigator will present the results of the heart from the CT scan. This will help us understand how best to explain the results of the CT scan to patients.

DETAILED DESCRIPTION:
This is a sub-study of the SCOT-HEART 2 trial (which aims to determine the best way to prevent heart attacks).

The purpose of this sub-study is to determine the effect of getting information on heart disease risk on lifestyle. At present doctors usually use a "risk score" to identify people at risk of heart disease who may benefit from medical treatment. In the SCOT-HEART 2 study the investigator will compare this "risk score" to a specialised heart scan (a computed tomography coronary angiogram or CTCA scan). In this study the investigator would like to understand more about the effects of receiving this information about the heart on lifestyle, including effects on smoking, diet and activity.

This study will recruit 400 participants who are taking part in the SCOT-HEART 2 trial. The investigator will assess lifestyle by using a detailed questionnaire which will be done at the start of the study and 6 months later. The investigator will also perform some simple investigations including a carbon monoxide breath test, blood pressure tests and measurements of activity such as step counts. This will help us understand the effects on lifestyle of getting information about a "risk score" or having a CT scan. In addition, for people who have CT scans the investigator will either provide a verbal explanation of the results, as is usual, or show pictures of the heart from the CT scan. This will help us understand how best to explain the results of the CT scan to partipants.

ELIGIBILITY:
Inclusion Criteria:

* MUST BE ENROLLED IN SCOTHEART 2 TRIAL

Exclusion Criteria:

* MUST BE ENROLLED IN SCOTHEART 2 TRIAL

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who meet National Institute for Heath and Care Excellence (NICE) recommendations on risk factor modifications | 6 months
  The primary endpoint will be the proportion of patients who meet NICE recommendations on diet, smoking, weight and activity levels (%)

SECONDARY OUTCOMES:
Smoking cessation | 6 months
  Proportion of patients who changed smoking habits (%)
Weight loss | 6 months
  Measure change in weight via body mass index and waist circumference (%)
Blood pressure control | 6 months
  Change in blood pressure control through lifestyle/compliance with medications (%)
Lipid levels | 6 months
  Change in serum lipid levels through lifestyle/compliace with medications (%)
Diabetic control | 6 months
  Change in glycosylated haemoglobin (HbA1c) (%)
Adherence to medications | 6 months
  Change in compliance with medications tracked through questionnaire
Exercise | 6 months
  Change in activity levels measured through activity monitoring (step count over 2 weeks) and international physical activity questionnaire
Quality of life/Anxiety and Depression | 6 months
  Change in quality of life measured through PHQ-9 (patient health questionnaire): anxiety and depression score (%)
ASSIGN score | 6 months
  Change in ASSIGN score as a result of lifestyle / risk factor modification (%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be made available to other researchers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: To be determined